CLINICAL TRIAL: NCT01670006
Title: Implantation of the Cochlear® Nucleus® System in Adults With Single-Sided Deafness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5397
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Single Sided Deafness
Keywords: Single sided deafness; Unilateral deafness; Unilateral hearing loss; Cochlear implantation
MeSH Terms: conditions — Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Cochlear Implantation (Experimental): Cochlear Nucleus Cochlear Implant System
  Interventions: Device: Cochlear Nucleus Cochlear Implant System

INTERVENTIONS:
Device: Cochlear Nucleus Cochlear Implant System

SUMMARY:
The objective of this feasibility study is to obtain preliminary safety and efficacy data associated with cochlear implantation in individuals with severe to profound sensorineural hearing loss contralateral to an ear with normal, or near-normal, hearing. The hypothesis is that restoration of hearing in the deafened ear will result in improved speech perception in the treated ear and advantages related to restoration of hearing to both ears.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Eighteen years-of-age or older at the time of implantation.
3. Presence of single-sided deafness as follows:

   1. Poorer ear (ear to be implanted):

      * severe to profound sensorineural hearing loss, defined as pure-tone thresholds 80 dB HL or greater for the frequencies 500, 1000, 2000, 3000, and 4000 Hz.
      * Monosyllabic word understanding, as measured using the CNC Word Test at 60 dBA under earphones, less than or equal to 10%.
   2. Better ear (contralateral ear):

      * Normal or near-normal hearing, defined as pure-tone thresholds no poorer than 30 dB HL at 250, 500, 1000, 2000, and 3000 Hz and no poorer than 40 dB HL at 4000 Hz.
      * Monosyllabic word understanding, as measured using the CNC Word Test at 60 dBA under earphones, of greater than or equal to 90%.
4. Duration of severe to profound sensorineural hearing loss of at least 6 months (to ensure stability of hearing loss) but no greater than 10 years.
5. English spoken as a primary language.

Exclusion Criteria:

1. Alleviation of tinnitus as the stated primary or sole motivation for seeking implantation by the subject and/or investigator.
2. Actively using an implantable device in the poorer ear.
3. Onset of severe to profound hearing loss < 6 years-of-age.
4. Evidence of active middle-ear pathology based on otologic examination and/or immittance testing.
5. Medical or psychological conditions that contraindicate undergoing surgery.
6. Ossification or any other cochlear anomaly at the implant ear that might prevent complete insertion of the electrode array.
7. Hearing loss of neural or central origin, including auditory neuropathy.
8. Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations inherent to the surgical procedure and prosthetic device.
9. Unwillingness and/or inability of the candidate to comply with all investigational requirements including, but not limited to, study protocol and surgical procedure, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Single-Sided Deafness and a Cochlear Implant: Ten subjects with Single-Sided Deafness (SSD) were implanted with a Cochlear Nucleus Cochlear Implant System and followed for 12 months after device activation.
Period: Overall Study
Arm/Group | Subjects With Single-Sided Deafness and a Cochlear Implant
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Single-Sided Deafness and a Cochlear Implant
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Device and procedure-related anticipated and unanticipated aderse events.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Subjects With Single-Sided Deafness and a Cochlear Implant
Number analyzed (Participants) | 10
participants | 1

2. Secondary Outcome: Hearing in Noise Test (HINT)Score
Description: To access speech perception performance using Hearing in noise test sentences in noise was measured at 12 months post activation. Recorded HINT sentences were presented to participants at 60dBA pre-operatively and 12 months post activation. Resultant score is percentage of words repeated correctly. Possible scores ranges from 0% to 100% correctly repeated. Higher percentage score means better outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of correct words.
Arm/Group | Subjects With Single-Sided Deafness and a Cochlear Implant
Number analyzed (Participants) | 10
percentage of correct words. | 10.9 (3.8)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Suspected allergic response to a drug used during the anesthesia procedure.
Arm/Group | Subjects With Single-Sided Deafness and a Cochlear Implant
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Single-Sided Deafness and a Cochlear Implant (N=10)
Sudden ventilation restriction upon induction of anesthesia (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other